CLINICAL TRIAL: NCT02694224
Title: A Randomized Phase II Pilot Study to Evaluate Safety and Efficacy of the Addition of Vismodegib to Standard Neoadjuvant Chemotherapy in Triple Negative Breast Cancer Patients
Brief Title: Addition of Vismodegib to Neoadjuvant Chemotherapy in Triple Negative Breast Cancer Patients
Acronym: SHH-CM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHH (Sonic HedgeHog)-CM
Record Dates: First submitted 2016-01-12; First posted 2016-02-29 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; triple negative; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — HhAntag691; Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vismodegib plus chemotherapy (Experimental): Vismodegib 150 mg orally during paclitaxel and then dose dense epirubicin + cyclophosphamide (EC) therapy (see active comparator arm)
  Interventions: Drug: vismodegib; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide
- chemotherapy (Active Comparator): Paclitaxel 80 mg/m2 weekly on days 1, 8 and 15 each 21 days x 12 doses and then dose dense E (90 mg/m2) plus cyclophosphamide (CPA) 600 mg/m2 each 2 weeks x 4 doses
  Interventions: Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: vismodegib — Smo inhibitor
  Other Names: GDC0449
  Arms: vismodegib plus chemotherapy
Drug: Paclitaxel — Paclitaxel (80 mg/m2) weekly x 12 doses followed by sequential dose dense Epirubicin (90 mg/m2) plus Cyclophosphamide (600 mg/m2) each 2 weeks x 4 doses with granulocyte macrophage colony stimulating factors (GM-CSF) support
Drug: Epirubicin — dose dense Epirubicin (90 mg/m2) plus Cyclophosphamide each 2 weeks x 4 doses with GMCSF after Paclitaxel
Drug: Cyclophosphamide — dose dense Cyclophosphamide (600 mg/m2) together with Epirubicin each 2 weeks x 4 doses with GMCSF after Paclitaxel

SUMMARY:
To evaluate safety and efficacy of vismodegib with standard neoadjuvant chemotherapy in breast cancer patients based on the CTCAE v4 2010

1. To study changes in biomarkers involved in the Hedgehog (HH) pathway in the first biopsy as compared to the later one
2. To detect predictive factors among patients who reached pathological complete response (pCR) as compared to those with no pCR
3. To evaluate the role of the addition of vismodegib in the pCR rate
4. To evaluate clinical responses by breast MRI and rates of breast conservative surgery after neoadjuvant chemotherapy
5. To evaluate QOL with EORTC QLQ-C30 scale

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Ability to give informed agreement and to carry out the whole study protocol during the study period
3. The patient should be able to carry out the needs of the clinical trial and have measurable disease
4. The patient should be 18-75 year-old
5. Triple negative breast cancer (ER<1%, Progesteron Receptor (PR)<1%, non-overexpressing HER2). 1. Patients with oligometastatic disease (1-2 resectable metastases) could be included
6. No previous systemic therapies
7. Patients who are going to benefit from neoadjuvant chemotherapy
8. Eastern Cooperative Oncology Group (ECOG)<2 or Karnofsky≥70%
9. Blood tests and biochemistry suitable: (absolute neutrophil count> 1500/uL; haemoglobin>9 gr/dL; platelets>100000/uL (microliters); total bilirubin≤ 1.5 the upper normal limit; GOT and GPT (transaminases)≤twice the upper normal limit; fasting glucose≤150 gr/dL; HbA1c≤8%, serum creatinine≤2 mg/dL.

Exclusion Criteria:

1. Severe diseases or infectious diseases or liver, kidney or bone marrow failure that advise not to participate in the study according to investigator criteria
2. Pregnancy or breast feeding period or fertility women who are not agree with contraception methods
3. Other primary tumors except for breast in situ carcinoma (CIS), cervical neoplasia(CIN) or localized skin tumors
4. Inflammatory breast cancer or bilateral breast cancer
5. Bone fractures, peptic ulcus or healing disorders
6. Any local or systemic therapy for breast cancer
7. To be maintained on immunosuppressants (prednisone > 10 mgr daily or others), aspirin> 325 mgr per day or clopidogrel > 75 mgr daily
8. Cardiomyopathy by New York Heart Association (NYHA) class II-IV; heart stroke in the previous 6 months; uncontrolled blood pressure (systolic > 150 mm Hg and /or diastolic > 100 mm Hg), coagulopathy or hemorrhagic diseases
9. Previous lung diseases
10. Personal history of abdominal perforation, abdominal abscess, or abdominal fistula.
11. Inability to swallow pills
12. Intolerance to galactose, malabsorption to galactose or/and glucose, or primary hypolactasia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | 21 months

SECONDARY OUTCOMES:
Molecular changes in breast | 30 months
Pathologic complete response (pCR) | 30 months
Clinical complete response (cCR) | 21 months
European Organisation for Research and Treatment of Cancer Quality of Life questionnaire C30 (EORTC QOL-C30) | 30 months
  We will consider data related to quality of life such as weakness, appetite, physical health, physiological health, social relationships, environment etc

CONTACTS AND LOCATIONS:
Overall Officials: Santisteban Marta, Doctor, Principal Investigator — Staff of the department of Oncology
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain